CLINICAL TRIAL: NCT00470535
Title: Phase II Study of Erlotinib (Tarceva®) in Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: Erlotinib in Treating Patients With Stage III or Stage IV Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated earlier due to a phase III study that showed this drug inferior to sorafenib
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000543406; RPCI-I-87106
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 - Oral Erlotinib hydrochloride (Experimental): Patients receive oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: erlotinib hydrochloride; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Oral
Other: immunohistochemistry staining method — Correlative Study
Other: laboratory biomarker analysis — Correlative Study

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with stage III or stage IV pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival (PFS) of patients with stage III or IV adenocarcinoma of the pancreas treated with erlotinib hydrochloride as first- or second-line therapy.

Secondary

* Determine the proportion of patients with a radiological response to this drug.
* Determine the overall survival of these patients.
* Determine the effect of this drug on quality of life in these patients.
* Correlate expression of EGFR, E-cadherin, P-cadherin, vimentin, cytokeratin, fibronectin, and ki67 in baseline tumor blocks and presence of K-ras mutations in baseline tumor biopsy specimens with response to this drug.
* Correlate smoking status with PFS in patients treated with this drug.
* Collect serum samples before, during, and after therapy for future serum proteomic studies and for development of profiles of responders to this drug.

OUTLINE: Patients receive oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

Patients complete a questionnaire about their smoking status at baseline. Patients also complete questionnaires about their quality of life every three weeks during study therapy and after completion of study therapy.

Blood samples are collected from patients at baseline and periodically during study for future serum proteomic research and for development of profiles of responders to erlotinib hydrochloride therapy. Paraffin-embedded tumor tissue from diagnostic tumor biopsies is assessed at baseline for expression of EGFR, E-cadherin, P-cadherin, vimentin, cytokeratin, fibronectin, and ki67 by immunohistochemical analysis. Tissue from surgical specimens in patients with prior resection is assessed for K-ras mutations by K-ras analysis.

After completion of study therapy, patients are followed for at least 6 months.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced inoperable or metastatic disease (stage III or IV disease)
* No more than 1 prior systemic therapy
* Patients who have not received 1 prior systemic therapy must meet 1 of the following criteria:

  * Ineligible for or refused chemoradiotherapy AND has stage III disease
  * Ineligible for or refused gemcitabine hydrochloride-based chemotherapy AND has stage IV disease
* No brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* WBC > 3,000/mm³
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN in patients with documented liver metastases)
* Creatinine < 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* No uncontrolled comorbid illness that is likely to increase toxicity of the study drug or to interfere with toxicity evaluation
* No known allergy to the study drug or its excipients
* No symptomatic interstitial pulmonary disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior adjuvant therapy allowed provided it was completed at least 28 days prior to study entry
* No prior EGFR-inhibitor
* No concurrent drugs that are known to be strong inducers or inhibitors of the CYP450 enzyme system
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent investigational or commercial agents or therapies with the intent to treat the patient's malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib (Tarceva): Erlotinib 150mg orally daily for three weeks
Period: Overall Study
Arm/Group | Erlotinib (Tarceva)
Started | 18
Completed | 0
Not Completed | 18
Not completed — Disease Progression | 13
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (10.2)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesion
Time Frame: Every cycle for up to 52 weeks
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 18
months | 1.4 [1.2 to 1.4]

2. Secondary Outcome: Clinical Response (Complete and Partial Response) as Measured by RECIST Criteria
Time Frame: After every cycle
Population: This study was terminated earlier due to a phase III study that showed this drug was not better than sorafenib so it didn't make sense to offer an inferior drug to patients.
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Overall Survival
Time Frame: After every cycle
Population: as for outcome 2
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Quality of Life (QOL) as Measured by EORTC PAN26 Every 3 Weeks During Study Therapy and After Completion of Study Therapy
Time Frame: Every 3 weeks
Population: as for outcome 2
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation of Smoking Status With Overall Survival
Time Frame: Every 3 weeks
Population: as for outcome 2
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation of Response, QOL, and Survival With EGFR, E-cadherin, P-cadherin, Vimentin, Cytokeratin, ki67, and Fibronectin and With Other Prognostic Variables, Such as Age and Tumor Grade
Time Frame: At Baseline
Population: as for outcome 2
Arm/Group | Erlotinib (Tarceva)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Erlotinib (Tarceva)
Serious Adverse Events (participants affected / at risk) | 9/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (Tarceva) (N=18)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 4 (4)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Blood glucose (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (Tarceva) (N=18)
Anaemia (Blood and lymphatic system disorders) | 9 (17)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 8 (12)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 12 (16)
Influenza like illness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 5 (5)
Pain (General disorders) | 2 (3)
Cholangiolitis (Hepatobiliary disorders) | 1 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (6)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5)
Alanine aminotransferase (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5)
Aspartate aminotransferase (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 8 (13)
Blood alkaline phosphatase (Investigations) | 8 (12)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood creatinine (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Prothrombin level abnormal (Investigations) | 1 (2)
Weight decreased (Investigations) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 5 (6)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (24)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 5 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (18)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated earlier due to a phase III study that showed this drug was not better than sorafenib

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes